CLINICAL TRIAL: NCT06010823
Title: A Prospective, Randomized, Open-label, Two-arms, Multi Center Feasibility Study to Evaluate the Safety and Efficacy of the PlaXtreme Device for Rehabilitation of the Hand in Post-stroke and Post TBI Participants
Brief Title: Safety and Efficacy Evaluation of the Robotic Enhanced Error Training of Upper Limb Function in Post-stroke and Post TBI Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reuth Rehabilitation Hospital (Other)
Collaborators: Loewenstein Hospital (Other); BioXtreme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0013-22-RRH
Record Dates: First submitted 2023-08-20; First posted 2023-08-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Brain Injuries; Paresis; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases
Keywords: Brain plasticity; Upper limb function; Robotic rehabilitation; Error augmentation or enhancement
MeSH Terms: conditions — Stroke; Brain Injuries; Paresis; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All the participants allocated to this group will undergo rehabilitation according to each medical center's standard rehabilitation practice. In addition, the participants will receive 12 therapy sessions incorporating error enhancement (3 session a week, for a period of 4 weeks), lasting approximately 25-30 minutes each.
  Interventions: Device: PlaXtreme
- Control (No Intervention): All participants allocated to this study group will undergo rehabilitation according to each medical center's standard rehabilitation practice.

INTERVENTIONS:
Device: PlaXtreme — A robotic device capable of applying motor error enhancement forces during upper limb practice in a virtual environment. The forces stimulate the body's instinctive adaptive response, which does not require the use of cognition to correct the patients hand movement.
  The device consists of a controller and specifically designed games projected on a screen requiring 3D active reaching movements. During the treatment sessions, the device will be operated by a trained occupational therapist.
  Arms: Intervention

SUMMARY:
Background: Cerebrovascular accident [CVA or commonly known as stroke] and traumatic brain injury (TBI) are common causes of morbidity, and motor impairments. Many stroke and TBI patients encounter severe functional impairments of their arm and/or hand. Recent studies have indicated that robotic training can improve upper limb function by enabling repetitive, adaptive, and intensive training.

One type of robotic training is error enhancement during three-dimensional movements. The goal of this approach is to elicit better accuracy, stability, fluidity and range of motion during reaching.

Previous research indicated the potential of robotic training with error enhancement as a viable clinical intervention for individuals facing motor deficits.

Objectives: To evaluate the safety and efficacy of a new robotic system based on error enhancement and intended for rehabilitation of motor hand functions of post-stroke and TBI patients.

Methods: A randomized, multi-center study with an open-label design. The study sample will consist of 96 participants who will be randomized into 2 separate groups. The intervention group consisting of 48 patients will receive training with the new robotic system, while the control group consisting of additional 48 patients will receive only standard practice treatments (with no exposure to the new robotic system). The outcomes of safety (adverse events and treatment tolerability), and efficacy (motor function, speed, tone, and spasticity) will be assessed and compared between the two groups. The assessment of the outcomes will be conducted at four different time points: (1) prior to the initiation of the four-week intervention, (2) after 2 weeks of intervention, (3) at the conclusion of the intervention, and (4) at a three-month follow-up session.

DETAILED DESCRIPTION:
Background: Stroke and traumatic brain injury (TBI) are leading causes for morbidity, hospitalization, and extended injury of motor system as well as movement learning. It has been proven that roughly 85% of stroke survivors suffer from weakness in their upper limbs, and around 40% of stroke survivors will suffer from severe handicap in their paretic arm, negatively affecting their independence and quality of life. Statically, about 50% - 70% of survivors will recover enough to enable daily use of their arm. These numbers indicate that although rehabilitation for stroke patients is evident, there remains a need for more effective methods.

Traditional rehabilitative methods are often time-consuming and labor-intensive. Only a few of these methods induce slightly improved arm function, and a full recovery is often not achieved. Recently, studies have indicated that robotic training has promise for improving functional abilities among stroke survivors by enabling repetitive, adaptive, intensive, and accurate control of task complexity during the rehabilitation period. One type of robotic training that is particularly promising is error enhancement; this utilizes the adaptive capabilities of the nervous system to improve fine motor function of the arm.

Study Objectives: To evaluate the change in the upper limb function amongst post-stroke and post-TBI patients undergoing error enhancement treatment compared to a control group in the following domains:

1. Motor Function (Fugl-Meyer Assessment, Action Research Arm Test (ARAT), pinch and grip tests)
2. Speed (Box and Blocks Assessment)
3. Tone and Spasticity (Modified Ashworth Scale)

In addition, this study will examine the safety and patient tolerability of the device.

Methods Population: A total of 96 participants will be recruited within 3 medical centers participating in the study. The recruitment will take place between 14 days and up to 18 months after the onset of the stroke or brain injury.

Recruitment: Electronic medical records of newly hospitalized patients will be screened to identify potential study participants. All eligible patients will be offered to participate. After obtaining informed consent, an intake session will take place for screening and evaluation purposes, conducted by a qualified occupational therapist. Patients successfully passing the screening session will undergo randomization to one of the two study arms with 1:1 ratio in each of the medical centers conducting the study.

All the treatments will be conducted a separate occupational therapist who will be blinded to the patient allocation group. Patients in the intervention arm will undergo training sessions with the robotic device, 3 times a week for a period up to 4 weeks, while the patients in the control arm will receive standard rehabilitative care.

Patients in both groups will undergo additional evaluation sessions at the following time points: after 2 weeks of intervention, at the conclusion of the intervention (4 weeks), and at a three-month follow-up session.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis due to first stroke (ischemic or hemorrhagic) or TBI;
* At least 14 days after the stroke or brain injury onset;
* No more than 18 months after stroke or brain injury onset;
* At least 4 weeks of remaining hospitalization in inpatient or outpatient rehabilitation ward;
* Voluntary provided informed consent obtained prior to any screening procedures;
* Cognitive status: Montreal Cognitive Assessment (MoCA test) score ≥ 22 or Mini Mental State Examination (MMSE) score > 24;
* Upper extremity function: Score between 35 and 52 points out of 66 on the Fugl- Meyer (FG) test with sub scores of 21-32/36 for the upper arm and 14-20/24 for the wrist and hand.

Exclusion Criteria:

* Complete paralysis of the affected side;
* Uncontrolled epilepsy;
* Upper-limb pain > 6 on 10-point Visual Analogue Scale (VAS);
* Concomitant or past medical conditions that might interfere with the study (i.e. hemi spatial neglect, orthopedic problems, etc.);
* Current participation in other interventional clinical study;
* Fingers spasticity score on the affected hand > 3 on Modified Ashworth Scale (MAS);
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ARAT score | 4 months
  The Action Research Arm Test (ARAT) is a reliable, valid and standardized assessment of post-stroke hemiparetic Upper Extremity functional limitations.
  The instrument contains 19 items grouped into 4 subtests; grasp, grip, pinch, and gross motor.
  Each item performance is rated on a 4-point scale (0=unable; 1=partial; 2= abnormal; 3=normal) and then item ratings are summed and reported out of 57 points with higher score indicating greater Upper Extremity function.
  In this study, the ARAT will be conducted only on the paretic hand.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | 4 months
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick and simple test, extensively used among a wide range of populations, including patients who have suffered from a stroke.
  During the assessment, the subject sits at a table in front of a box with two compartments. The first has 150 blocks, while the second is empty. The participant must move as many blocks as he or she can (one at a time) in 60 seconds. The final score is the number of moved blocks out of a possible score of 150.
  During the assessment, the box should be oriented lengthwise and placed at the client's midline, with the compartment holding the blocks oriented towards the hand being tested. In order to practice and register baseline scores, the test should begin with the unaffected upper limb. Additionally, a 15-second trial period is permitted at the beginning of each side.
  In this study, the BBT will be conducted on both of the patient's hands.
Pinch test | 4 months
  The Pinch test evaluates hand and upper extremity. The measurements are conducted using a pinch dynamometer by squeezing the pinch meter between the thumb and forefinger.
  In this study, the Pinch test will be conducted on both of the patient's hands.
Fugl-Meyer Assessment | 4 months
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. Scale items are scored on the basis of ability to complete each item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226. This FMA score for a paretic upper limb may range from 0 to 66, with a lower score indicating higher impairment. The FMA scores will be used in this study not only for evaluation, but also as an inclusion criterion, as described in the inclusion/exclusion criteria section.
Functional Ambulatory Category | 4 months
  Functional Ambulation Categories (FAC) classify the patient's walking as dependent or non-dependent. This is a visual measurement of walking scored according to 6-point scale to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
  * A score of 0 indicates that the patient is a non-functional ambulator (cannot walk);
  * A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3)
  * A score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score)
Trunk control test | 4 months
  The Trunk Control Test (TCT) is used to assess trunk movements in patients that have suffered from a neurological disorder (i.e stroke) The test consists of four tasks performed on a bed: rolling to a weak side, rolling to a strong side, balance in sitting position on the edge of the bed with the feet off the ground for at least 30 seconds and sitting up from a lying down position. Each task is graded with the following scores: 0 = for inability to perform the task, 12= if subject is able to perform the task but with help or in an abnormal style and 25=if subjects is able to perform the task normally. The total score ranges from 0 to 100 points, with higher score indicating better performance.
Modified Ashworth Scale | 4 months
  The Modified Ashworth Scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform. It is performed by extending the patient's limb from a position of maximal possible flexion to maximal possible extension. Afterwards, the patient is assessed while moving from extension to flexion.
  In this study, the MAS will be conducted only on the paretic hand.
Visual Analogue Scale (VAS) | 4 months
  The Visual Analogue Scale is a pain rating scale used to determine pain severity and intensity. A standard analog scale ranges (0) meaning no pain to (10) meaning the worst pain imaginable. A patient has to mark a point on the line that matches the amount of pain he or she are experiencing.
Grip test | 4 months
  The grip test using dynamometer assesses the maximum grip force to evaluate the grip strengh of the hand.
Clinical Global Impression Scale (CGI) | 4 months
  Clinical Global Impression Scale (CGI) severity is a 3-item observer-rated scale that measures illness severity (CGIS), global improvement or change (CGIC) and therapeutic response. The assessdment tool provided with a seven-point scale of severity of patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Mansour, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (2):
- Israel (2):
  - Loewenstein Rehabilitation Center, Raanana
  - Reuth Rehabilitation Hospital, Tel Aviv